CLINICAL TRIAL: NCT04999917
Title: High-resolution PET-CT Imaging for Intraoperative Margin Assessment in Early-stage Breast Cancer: a Prospective Multicentric Interventional Clinical Study
Brief Title: Specimen PET-CT Imaging for Intraoperative Margin Assessment in Breast Cancer
Acronym: BrIMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: XEOS Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BrIMA
Record Dates: First submitted 2021-08-02; First posted 2021-08-11 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Breast Cancer Invasive; Breast Cancer in Situ
Keywords: PET-CT; margin assessment; breast conserving surgery
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intraoperative high-resolution PET-CT imaging of resected breast tumor. (Experimental)
  Interventions: Diagnostic Test: high-resolution PET-CT specimen imaging.

INTERVENTIONS:
Diagnostic Test: high-resolution PET-CT specimen imaging. — A single intravenous injection of 18F-FDG (0.80 MBq/kg) is given between 30 minutes and 3 hours before tumor resection.
  Surgical resection of the breast tumor (= main specimen) under general anesthesia.
  The main specimen is imaged using the Aura 10 PET-CT Specimen Imager (XEOS Medical, Ghent, Belgium). In case of positive margins, the surgeon will perform oriented cavity shaving. The cavity shaves and lymph nodes (if any) are also imaged using the Aura 10 PET-CT Specimen Imager (for scientific purposes only).
  The main specimen and if applicable the cavity shaves and lymph node(s) are processed following standard-of-care routine: from tissue samples to HE-stained and IHC-stained sections. The histopathological margin status shall be reported according to the ASCO-CAP guidelines, and shall be compared to the PET-CT images of the resected specimens.

SUMMARY:
Breast-conserving surgery (BCS) has become the standard-of-care for surgical management of the majority of women with early-stage breast cancer. Successful BCS entails excision of the tumor with an adequate amount of surrounding healthy breast parenchyma, such that negative resection margins are obtained. Despite efforts to obtain tumor-free margins, approximately 20-30% of women still require reoperation.

The rationale of this study is to examine the contribution of the adjunctive use of perioperative high-resolution PET-CT specimen imaging in early-stage breast cancer to the identification of all positive resection margins during breast-conserving surgery. Histopathological findings of the breast tumor specimen are applied as the gold standard.

After a successful screening phase and after informed consent is provided, the patient will enroll the study. The preparations for the BCS proceed following the routine protocol (i.e. as if the patient would not participate in the study). In addition to these standard preparations, on the day of surgery the patient will receive a study-specific injection with a low dose of a radiotracer substance (18F-FDG; 0.8 MBq/kg). Before injection, the blood sugar level will be measured by a small finger prick. If the blood sugar level is good, the radiotracer substance will be intravenously administered. The injection is given at the nuclear medicine department between 30 minutes and 3 hours before surgery. After the injection was given, the patient will be transferred to the operating theatre. The breast tumor will be removed in the same way as if the patient is not participating in the study. As soon as the tumor is excised, it will be imaged using the specimen PET-CT scanner in the operating theatre. While waiting for these 3D images, the surgeon will remove the lymph nodes, if applicable. The breast surgeon will then evaluate the 3D images of the removed breast tumor. In case of suspected positive margins, the surgeon will excise additional breast tissue to ensure that all tumor tissue is excised during this surgery. For scientific purposes only and if available, the cavity shaves and resected lymph nodes will also be imaged with the specimen PET-CT scanner. No clinical decisions that could affect further treatment will be based on this. After surgery, all excised tissues will be sent to the pathology department. This is standard routine and is also done for patients not participating in the study. A routine follow-up visit will be planned with the surgeon. During that routine visit, a staff member of the study team will ask additional study-related questions regarding possible complications. If the latter is not possible during the standard follow-up visit, a staff member of the study team will contact the patient by phone call 1-3 weeks after surgery. The study is completed after this follow-up visit or phone call.

ELIGIBILITY:
Inclusion Criteria:

* females with an age over 18 years;
* confirmed breast cancer (IDC, DCIS, ILC) with indication to undergo BCS;
* a minimal tumor size of 1.0 cm (in at least one dimension):

  * IDC group: assessed preoperatively on ultrasound;
  * DCIS subgroup: assessed preoperatively on mammogram;
  * ILC subgroup: assessed preoperatively on ultrasound;
  * NAT subgroup: assessed after NAT and before surgery on ultrasound;
* patients with IDC who have received NAT (i.e. chemotherapy, immunotherapy or endocrine therapy until eight weeks before BCS) may participate in the study;
* vacuum-assisted core breast biopsy is allowed in the DCIS subgroup only;
* able to understand treatment protocol and informed consent form;
* estimated by the investigator to be compliant for study participation.

Exclusion Criteria:

* general or local contra-indication for BCS;
* previous breast surgery;
* inflammatory breast cancer;
* radiotherapy of the ipsilateral breast;
* vacuum-assisted core breast biopsy for all patients allocated to the IDC, ILC or NAT subgroup (vacuum-assisted core breast biopsy is allowed in the DCIS subgroup as long as the residual tumor size on mammogram is at least 1.0 cm);
* patients with DCIS only or ILC, and that have received NAT;
* blood glucose level over 200 mg/dL on the day of surgery;
* pregnancy or lactation;
* participation in other clinical studies with a radiation exposure of more than 1 mSv in the past year;
* active bacterial, viral or fungal infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Perioperative addressing positive margins of the invasive component in IDC. | Perioperative (day 0).
  The primary effectiveness endpoint is a measure of perioperative success in addressing positive margins of the invasive component with the adjunctive use of high-resolution PET-CT specimen imaging as detected by permanent pathology in the IDC subgroup.

SECONDARY OUTCOMES:
Perioperative addressing positive margins of the invasive component in breast cancer. | Perioperative (day 0).
  A measure of perioperative success in addressing positive margins of the invasive component with the adjunctive use of high-resolution PET-CT specimen imaging as detected by permanent pathology in:
  * the total study population excluding the DCIS subgroup (IDC + ILC + NAT);
  * the ILC subgroup;
  * the NAT subgroup.
Perioperative addressing any positive margin in breast cancer. | Perioperative (day 0).
  A measure of perioperative success in addressing any positive margin with the adjunctive use of high-resolution PET-CT specimen imaging as detected by permanent pathology in:
  * the total study population (IDC + DCIS + ILC + NAT);
  * the IDC subgroup;
  * the DCIS subgroup;
  * the ILC subgroup;
  * the NAT subgroup.
Perioperative success in obtaining final negative margins of the invasive component in breast cancer. | Perioperative (day 0).
  A measure of perioperative success in obtaining final negative margins of the invasive component as detected by permanent pathology (1) by the additional use of high-resolution PET-CT imaging and (2) by additional use of standard-of-care in:
  * the total study population excluding DCIS (IDC + ILC + NAT);
  * the IDC subgroup;
  * the ILC subgroup;
  * the NAT subgroup.
Perioperative success in obtaining final negative margins in breast cancer. | Perioperative (day 0).
  A measure of perioperative success in obtaining final negative margins (invasive and/or in situ component) as detected by permanent pathology (1) by the additional use of high-resolution PET-CT imaging and (2) by additional use of standard-of-care in:
  * the total study population (IDC + DCIS + ILC + NAT);
  * the IDC subgroup;
  * the DCIS subgroup;
  * the ILC subgroup;
  * the NAT subgroup.
Final positive margins of the invasive component after breast-conserving surgery. | Perioperative (day 0).
  A measure of the number of patients with final positive resection margins of the invasive component after BCS in:
  * the total study population excluding DCIS (IDC + ILC + NAT);
  * the IDC subgroup;
  * the ILC subgroup;
  * the NAT subgroup.
Final positive margins of any margin after breast-conserving surgery. | Perioperative (day 0).
  A measure of the number of patients with final positive resection margins (invasive and/or in situ component) after BCS in:
  * the total study population (IDC + DCIS + ILC + NAT);
  * the IDC subgroup;
  * the DCIS subgroup;
  * the ILC subgroup;
  * the NAT subgroup.
Diagnostic performance based on the invasive component of breast cancer. | Perioperative (day 0).
  Sensitivity, specificity, positive and negative predictive value, failure rate and, interobserver reproducibility of high-resolution PET-CT imaging based on the invasive component of:
  * the total study population excluding DCIS (IDC + ILC + NAT);
  * the IDC subgroup;
  * the ILC subgroup;
  * the NAT subgroup.
Diagnostic performance based on any margin of breast cancer. | Perioperative (day 0).
  Sensitivity, specificity, positive and negative predictive value, failure rate and, interobserver reproducibility of high-resolution PET-CT imaging based on any margin of:
  * the total study population (IDC + DCIS + ILC + NAT);
  * the IDC subgroup;
  * the DCIS subgroup;
  * the ILC subgroup;
  * the NAT subgroup.
Reoperation rate. | Follow-up visit (+/- week 2).
  The number of patients that require a second or a third surgery due to positive margins at initial primary breast-conserving surgery and the type of repeat surgery (BCS or mastectomy).
Resected tissue volume. | Perioperative (day 0).
  The volume (mm³) of resected main specimen, and possible cavity shaves after PET-CT imaging and possible cavity shaves after standard-of-care approach.
Detection of malignant cells in cavity shaves and resected lymph nodes. | Perioperative (day 0).
  A measure of success in detecting malignant cells in resected lymph nodes and cavity shaves with the adjunctive use of high-resolution PET-CT specimen imaging as detected by permanent pathology.

CONTACTS AND LOCATIONS:
Locations (1):
- Gynecology department, Ghent, Flanders, Belgium